CLINICAL TRIAL: NCT05451511
Title: Rapid Acceleration of Diagnostics Underserved Populations Supplement Rent Relief and COVID-19 in St. Louis: COVID-19 Resource Offers Among Rent and Utility Assistance Applicants in St. Louis
Brief Title: COVID-19 Resource Offers Among Rent and Utility Assistance Applicants in St. Louis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Matthew Kreuter, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3R01CA235773-03S2 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-07-11 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Behavior and Behavior Mechanisms; Communication
MeSH Terms: conditions — Behavior; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Door-In-The-Face Technique (Active Comparator): Using sequential request strategies, participants randomized to the Door-In-The-Face Technique group will be asked if they would like vaccination support (if not already vaccinated) and if they say no, they will be asked if they'd like to try a COVID-19 self-test at home.
  Interventions: Other: Door-In-The-Face Technique
- Foot-In-The-Door Technique (Active Comparator): Using sequential request strategies, participants randomized to the Foot-In-The-Door Technique group will be first asked if they are interested in trying an at-home COVID-19 test and then asked if they are interested in vaccination support (if not already vaccinated).
  Interventions: Other: Foot-In-The-Door Technique

INTERVENTIONS:
Other: Door-In-The-Face Technique — Sequential request strategies will be applied as an intervention. For the Door-In-The-Face Technique, participants first receive a large request they are unlikely to accept, followed by a smaller request that is the true behavior of interest.
  Arms: Door-In-The-Face Technique
Other: Foot-In-The-Door Technique — Sequential request strategies will be applied as an intervention. For the Foot-In-The-Door Technique, participants are shown an easier first request that they are likely to accept, followed by a larger request that is not the behavior of interest.
  Arms: Foot-In-The-Door Technique

SUMMARY:
The purpose of this study is to evaluate health messaging strategies that help individuals with a high degree of housing-related needs engage in COVID-19 vaccination and testing behaviors. Findings from this research can help other communities determine how best to integrate social needs and COVID-19 prevention services. Participants' contact information will be shared with us by 211 with the participants' previously given consent. The study team will send via text message a link to a survey that includes a screen where they will provide informed consent. Those who provide consent will be randomly assigned to receive one of two surveys. The order of the offers is what varies across the surveys. Participants will be asked, along with other survey items, if they have been vaccinated against COVID-19. If they have not, they will be asked if they are interested in receiving help to receive a vaccine. Participants will also be asked if they are interested in receiving an at-home COVID self-test. If they say yes to assistance with vaccination, a vaccine navigator will call and assist them. If they say yes to receiving a COVID test, the study team will ship them a test that has been procured from the City of St. Louis Mayor's office. One month later participants will be sent a follow-up survey that asks about their experiences either with testing or with vaccination if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Applicants for rent and utility assistance in St. Louis City or County
* English language proficiency
* Be willing to be contacted via text message or email
* Resident of St. Louis City or County

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Proportion Vaccinated | Baseline
  Via a mobile-optimized web-based survey, the investigators will ask individuals seeking rental/housing assistance if they are thinking about getting vaccinated and report the proportion "already vaccinated."
Sequential Request Strategy Effectiveness | Baseline
  To compare differences in testing acceptance and vaccination responses by sequential request strategy, the investigators will identify which strategy is associated with greater testing and vaccination intentions.
Testing and Vaccination Offer Acceptance | Baseline
  At baseline, participants will be offered vaccination support and free a COVID-19 self-test. The investigators will report the proportion of applicants who accept each of the offers.

SECONDARY OUTCOMES:
Testing and Vaccination Behaviors | 1 month follow-up
  After one month follow-up, the investigators will report the proportion of participants who complete the self-test and report the results, and report having been vaccinated since the baseline survey.
Rent Relief | Baseline
  The investigators will ask about the outcome of rent or utility assistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided